CLINICAL TRIAL: NCT02347267
Title: The Impact of Reduction in Consumption of Caloric and no Caloric Sweetened Beverages on Weight, Body Composition and Blood Pressure in Young Adults.
Brief Title: Reduction in Consumption of Sweetened Beverages on Weight, Body Composition and Blood Pressure in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, LILIA CASTILLO MARTINEz, at the National Institute of Medical Science and Nutrition Salvador Zubiran, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clic 002
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Obesity and Overweight
Keywords: Beverages sweetened caloric, no caloric; Weight; Fat percentage; Body Composition; Blood pressure; Sugar; Sodium; Dietary intake
MeSH Terms: conditions — Obesity; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Caloric and non-caloric SSBS reduction (Experimental): Sweetened beverages (SSBS) caloric and non-caloric were not permitted and allowed only plain water
  Interventions: Behavioral: Caloric and non-caloric SSBS reduction
- Caloric SSBS reduction (Active Comparator): Only plain water and non-caloric sweetened beverages (SSBS) were allowed
  Interventions: Behavioral: Caloric SSBS reduction
- All beverages (No Intervention): Beverages were not restricted

INTERVENTIONS:
Behavioral: Caloric and non-caloric SSBS reduction — Isocaloric individualized diet and sweetened caloric and non-caloric beverages restriction
  Arms: Caloric and non-caloric SSBS reduction
Behavioral: Caloric SSBS reduction — Isocaloric individualized diet and caloric SSBS restriction
  Arms: Caloric SSBS reduction

SUMMARY:
The impact of reduction in consumption of caloric and no caloric sweetened beverages on:

* weight
* body composition
* blood pressure
* young adults

DETAILED DESCRIPTION:
The number of overweight and obese individuals has recently increased considerably. The World Health Organization estimates that there are 1.4 billion overweight and obese people in the world (1); in Mexico alone 70% of the adult population suffers from overweight and obesity, and 34.4% of school age children are above their normal weight (2) At the same time, hypertension affects more than a third of adults throughout the world and contributes to 9.4 million deaths a year from heart disease (3). In Mexico there are 22.4 million adults with hypertension, only 5.7 of whom are controlled (4). Obesity and hypertension are associated with life style both in the world and in Mexico, where changes in eating habits with increased fat in the diet, overconsumption of soft drinks and refined sugars and decrease in physical activity have led to numerous diseases (4). Mexico is the Latin American country with the highest consumption of carbonated beverages (5), averaging 384 soft drinks/person/year (6). The diminished sensation of satiety and the high ingestion of simple sugars (7, 8) facilitate the formation of triglycerides stored in fatty tissue and overweight and obesity (9, 10). Recent studies have examined the relationship between beverages and weight, albeit with controversial results. The majority of the studies have focused on increased consumption of sweetened drinks and their effect on weight over short periods of time (11,13,14). Meanwhile, consumption of low calorie beverages has increased, although there is no consensus about the utility of substituting sugar with artificial sweeteners to achieve better weight control (13). As much as obesity is a world-wide health issue, it is important to establish whether beverages with artificial sweeteners can aid in regulating weight. Since soft drinks contain sodium, it is also important to determine whether elevated sodium ingestion from them could increase blood pressure. Recent studies have demonstrated an association between sugar sweetened beverages and blood pressure, but the majority have been observational (14) and have not analyzed all types of sweetened beverages (15, 16).Because of these issues, the objective of the present study was to characterize the effect of reducing the consumption of beverages with sugar and artificial sweeteners on weight and blood pressure on nursing students. The working hypothesis was that nursing students from the National Institute of Medical Science and Nutrition in Mexico City (INCMNSZ) who substituted their intake of sugar or artificially sweetened soft drinks with plain water would have greater weight loss, lower fat and lower blood pressure than students who did not diminish their intake of soft drinks.

ELIGIBILITY:
Inclusion Criteria:

Students in the Bachelor of Nursing INCMNSZ. What made light and moderate physical activity no more than 1 hour of exercise.

That according to the survey conducted consume at least one sugary drink according to the recommendations of the Ministry of Health

Exclusion Criteria:

Subjects who currently have or meet a specific diet. Diagnosed with hypertension or utilization of antihypertensive drugs. Hyperthyroidism and hypothyroidism. Use of drugs for weight loss. Diabetes mellitus History of cardiovascular events. Peripheral vascular disease. Cancer. Renal damage Psychiatric illness

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage of change from baseline in kilograms of weight | Baseline to three and six months

SECONDARY OUTCOMES:
Percentage of change from baseline in diastolic blood pressure | Baseline to three and six months follow-up
Percentage of change from baseline in systolic blood pressure | Baseline to three and six months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marisela Vázquez Duran, M.Sc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Lilia Castillo Martinez, M.Sc, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Arturo Orea Tejeda, M.D, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- INCMNSZ, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Rivera JA, Munoz-Hernandez O, Rosas-Peralta M, Aguilar-Salinas CA, Popkin BM, Willett WC; Comite de Expertos para las Recomendaciones. [Beverage consumption for a healthy life: recommendations for the Mexican population]. Salud Publica Mex. 2008 Mar-Apr;50(2):173-95. doi: 10.1590/s0036-36342008000200011. Spanish. PMID 18372998
- [Background] Bray GA, Nielsen SJ, Popkin BM. Consumption of high-fructose corn syrup in beverages may play a role in the epidemic of obesity. Am J Clin Nutr. 2004 Apr;79(4):537-43. doi: 10.1093/ajcn/79.4.537. PMID 15051594
- [Background] Ma J, Chang J, Checklin HL, Young RL, Jones KL, Horowitz M, Rayner CK. Effect of the artificial sweetener, sucralose, on small intestinal glucose absorption in healthy human subjects. Br J Nutr. 2010 Sep;104(6):803-6. doi: 10.1017/S0007114510001327. Epub 2010 Apr 27. PMID 20420761
- [Background] Gibson S. Sugar-sweetened soft drinks and obesity: a systematic review of the evidence from observational studies and interventions. Nutr Res Rev. 2008 Dec;21(2):134-47. doi: 10.1017/S0954422408110976. PMID 19087367
- [Background] Vartanian LR, Schwartz MB, Brownell KD. Effects of soft drink consumption on nutrition and health: a systematic review and meta-analysis. Am J Public Health. 2007 Apr;97(4):667-75. doi: 10.2105/AJPH.2005.083782. Epub 2007 Feb 28. PMID 17329656